CLINICAL TRIAL: NCT01919515
Title: Randomized Controlled Clinical Trial of a New NuSmile ZR Esthetic Primary Molar Crown
Brief Title: Trial of a New NuSmile ZR Esthetic Primary Molar Crown
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NuSmile, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130203
Record Dates: First submitted 2013-07-31; First posted 2013-08-09 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Dental Caries
Keywords: pediatric; primary molars; stainless steel crowns
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZR Crown & Stainless Steel Crown (Other): Each subject will have a maximum of one ZR Crown and one Stainless Steel Crown cemented on primary molars that are treatment planned for a crown.
  Interventions: Device: ZR Crown; Device: Stainless Steel Crown

INTERVENTIONS:
Device: ZR Crown — This is an esthetic primary molar crown.
Device: Stainless Steel Crown — This is a conventional stainless steel crown.

SUMMARY:
The hypothesis to be tested is that NuSmile ZR esthetic primary molar crowns perform similarly to an established Stainless Steel primary molar crown (3M ESPE) for restoration of primary molar teeth.

DETAILED DESCRIPTION:
The aim of this study is to clinically evaluate the performance of a new NuSmile ZR esthetic primary molar crown, compared with 3M ESPE Primary Stainless Steel crowns (currently the most common full coverage crown for the restoration of primary molars when a crown is necessary)in the restoration of 50 paired, prepared primary first and second molar teeth in the deciduous dentition of child patients.

ELIGIBILITY:
Inclusion Criteria:

* Be between 3 and 7 years of age
* Have a minimum of two primary molar teeth, requiring crowns
* Have a parent or guardian capable of giving written informed consent
* Have study teeth in occlusion and in contact with adjacent teeth
* Teeth to be included in the study must have adequate remaining tooth tissue for retention of the NuSmile ZR crown to allow randomization of treatments to teeth.

Exclusion Criteria:

* Tooth is considered to be within 36 months of exfoliation
* They have a severe / serious childhood illness that requires frequent hospitalization
* They have poor general health
* They have juvenile periodontitis
* Patient is unable to return for evaluations / study recalls

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Assessments of the SSC and ZR Crown | At Baseline
  Clinically evaluate both the stainless steel crown and ZR crown for wear, gingival health, crown performance, color match, marginal integrity.
Assessments of the SSC and ZR Crown at 6 months | 6 month visit
  Clinically evaluate both the stainless steel crown and ZR crown for wear, gingival health, crown performance, color match and marginal integrity.
Assessments of the SSC and ZR Crown at 12 months | 12 month visit
  Clinically evaluate both the stainless steel crown and ZR crown for wear, gingival health, crown performance, color match and marginal integrity.
Assessments of the SSC and ZR Crown at 18 months | 18 month visit
  Clinically evaluate both the stainless steel crown and ZR crown for wear, gingival health, crown performance, color match and marginal integrity.
Assessments of the SSC and ZR Crown at 24 months | 24 month visit
  Clinically evaluate both the stainless steel crown and ZR crown for wear, gingival health, crown performance, color match and marginal integrity.
Assessments of SSC and ZR Crown at 36 months | 36 month visit
  Clinically evaluate both the stainless steel crown and ZR crown for wear, gingival health, crown performance, color match and marginal integrity.
Assessments of SSC and ZR Crowns at 48 months | 48 month visit
  Clinically evaluate both the stainless steel crown and ZR crown for wear, gingival health, crown performance, color match and marginal integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J. Donly, D.D.S., M.S., Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - The University of Texas Health Science Center-Dental School, San Antonio, Texas
  - The University of Texas Health Science Center-Ricardo Salinas Dental Clinic, San Antonio, Texas

REFERENCES:
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Ryge G. Clinical criteria. Int Dent J. 1980 Dec;30(4):347-58. PMID 6935165